CLINICAL TRIAL: NCT01615120
Title: Phase II, Open Label Study of the Effect of GTx-758 as Secondary Hormonal Therapy on Serum PSA and Serum Free Testosterone Levels in Men With Metastatic Castration Resistant Prostate Cancer Maintained on Androgen Deprivation Therapy
Brief Title: Study of the Effect of GTx-758 on Serum PSA and Testosterone in Men With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GTx (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G200712
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Results first posted 2021-02-16 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 3-fluoro-N-(4-fluorophenyl)-4-hydroxy-N-(4-hydroxyphenyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GTx-758 125mg (Experimental): one GTx-758 tablet orally administered daily
  Interventions: Drug: GTx-758 125 mg
- GTx-758 250 mg (Experimental): two GTx-758 tablets orally administered daily
  Interventions: Drug: GTx-758 250 mg

INTERVENTIONS:
Drug: GTx-758 125 mg — One 125 mg tablet once a day
  Arms: GTx-758 125mg
Drug: GTx-758 250 mg — two 125 mg tablets once daily
  Arms: GTx-758 250 mg

SUMMARY:
Protocol G200712 is a Phase II, exploratory study to assess the effects of GTx-758 on serum prostate specific antigen (PSA) response ans serum PSA progression in men with Metastatic Castration Resistant Prostate Cancer (mCRPC) on Androgen Deprivation Therapy (ADT) with luteinizing hormone-releasing hormone (LHRH) agonists, LHRH antagonists, or orchidectomy. This study will also assess the venous thromboembolism (VTE) risk of lower doses of GTx-758.

ELIGIBILITY:
Inclusion Criteria:

* Be over age 18 years
* Be able to Communicate effectively with the study personnel
* Have histologically confirmed prostate cancer
* Have castration resistant prostate cancer patients with radiographic evidence of metastatic disease (T any - N any - MI)
* ECOG performance status of 0 to 2
* Have been treated with ADT (chemical or surgical) for at least 6 months
* Have a castrate level of serum total testosterone (< 50ng/dL)
* Have a history of serum PSA response on ADT. A serum PSA response is an undetectable level of serum PSA (≤ 0.2/mL) or at least a 90% reduction in serum PSA from the serum PSA value prior to the initiation of treatment to < 10ng/mL
* Have a rising serum PSA on two successive assessments at least 2 weeks apart and serum PSA levels ≥ 2ng/mL or > 2 ng/mL and a 25% increase above the nadir from the ADT.
* Be continued on ADT throughout this study
* give written informed consent prior to any study specific procedures
* subjects must agree, if not already on anticoagulation therapy or aspirin, to take 81 mg aspirin daily throughout the duration of their participation in this study and for 30 days after completion of dosing with GTx-758.
* Subjects must agree to use acceptable methods of contraception:
* If their female partners are pregnant or lactating, acceptable methods of contraception from the time of the first administration of study medication until 3 months following administration of the last dose of study medication must be used. Acceptable methods are: condom used with spermicidal foam/gel/film/cream/suppository. If the subject has undergone surgical sterilization (vasectomy with documentation of azospermia), a condom with spermicidal foam/gel/film/cream/suppository should be used.
* If the male subject's partner could become pregnant, use acceptable methods of contraception from the time of the first administration of study medication until 3 months following administration of the last dose of study medication.Acceptable methods of contraception are as follows: condom with spermicidal foam/gel/film/cream/suppository [i.e., barrier method of contraception], surgical sterilization (vasectomy with documentation of azospermia) and a barrier method {condom used with spermicidal foam/gel/fil/cream/suppository}, the female partner uses oral contraceptives (combination estrogen/progesterone pills), injectable progesterone or subdermal implants and a barrier method {condom used with spermicidal foam/gel/film/cream/suppository}.
* If the female partner has undergone documented tubal ligation (female sterilization), a barrier method {condom used with spermicidal foam/gel/film/cream/suppository} should be used
* If the female partner has undergone documented placement of an intrauterine device (IUD) or intrauterine system (IUS), a barrier method {condom with spermicidal foam/gel/film/cream/suppository} should also be used.

Exclusion Criteria:

* Known hypersensitivity or allergy to estrogen or estrogen like drugs
* Need for urgent chemotherapy, radiation therapy or surgical intervention for prostate cancer in the opinion of the investigator;
* Any disease or condition (medical or surgical) which might compromise the hematologic, cardiovascular, endocrine, pulmonary, renal, gastrointestinal, hepatic, or central nervous system; or other conditions that may interfere with the absorption, distribution, metabolism or excretion of study drug, or would place the subject at increased risk
* Subjects with a personal history of abnormal blood clotting or thrombotic disease (venous or arterial thrombotic events such as history of stroke, deep vein thrombosis (DVT), and or pulmonary embolus (PE)).
* Any subjects, as determined by a central laboratory, with

  1. a modified activated protein C reaction ratio ≤ 2.5 and a Factor V Leiden gene mutation,
  2. an antithrombin level below the lower limit of the normal range,
  3. an antiphospholipid antibody level that is indeterminate, positive, or outside the normal range,
  4. or a prothrombin gene mutation
* Symptomatic congestive heart failure (NYHA Class III - IV), unstable angina pectoris, cardiac arrhythmia, or history of atrial fibrillation
* The presence of consistently abnormal laboratory values which are considered clinically significant. In addition, any subject with liver enzymes (ALT or AST) above 2 times the upper limit of normal, total bilirubin above 2 times the upper limit of normal, or serum creatinine above 1.5 times the upper limit of normal will NOT be admitted to the study.
* Received an investigational drug within a period of 90 days prior to the enrollment in the study.
* Received the study medication GTx-758 previously;
* Currently taking testosterone, testosterone like agents, 5a-reductase inhibitor (finasteride, dutasteride),or antiandrogens (bicalutamide, flutamide or nilutamide). Subjects taking a 5a-reductase inhibitor or one of these antiandrogens may be eligible if the subject undergoes a 6 week washout period after stopping therapy. The subject must have at least two rising serum PSA levels at least 2 weeks apart after therapy with these 5a-reductase inhibitor or these antiandrogens have been stopped (antiandrogen withdrawal)and complete the 6-week washout period to be eligible;
* Have previously taken or are currently taking diethylstilbestrol, other estrogens, abiraterone or ketoconazole or any other inhibitor of CYP17 (17a-hydroxylase/C17,20-lyase);
* Currently having radiation therapy to prostate for cancer control (radiation to bone to relieve pain is acceptable)
* Have previously taken or are currently taking enzalutamide;
* Have previously received cytotoxic chemotherapy for prostate cancer;
* Recent hospitalization (within 30 days of screening);
* Recent surgery (within 30 days of screening);
* Have taken body building or fertility supplements within 4 weeks of admission into the study;
* Have been previously diagnosed or treated for active cancer (other than prostate cancer or non-melanoma skin cancer)within the previous five years;
* Have a BMI > 35.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2012-08-14 (Actual); Primary Completion 2016-11-09 (Actual); Study Completion 2016-11-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (26):
- United States (26):
  - Urology Associates Medical Group, Burbank, California
  - VA of Greater Los Angeles, Los Angeles, California
  - Tower Urology, Los Angeles, California
  - San Bernardino Urological Assoc., San Bernardino, California
  - Genesis Healthcare Partners, San Diego, California
  - Urology Specialists of So. California, Torrance, California
  - Univ. of Colorado Cancer Center, Aurora, Colorado
  - Connecticut Clinical Research Center, Middlebury, Connecticut
  - So. Florida Medical Research, Aventura, Florida
  - AMPM Research, Miami, Florida
  - Coastal Medical Center, Sarasota, Florida
  - GTx Investigative Site, St. Petersburg, Florida
  - Pinellas Urology, St. Petersburg, Florida
  - Urology of Indiana, Greenwood, Indiana
  - First Urology PSC, Jeffersonville, Indiana
  - Chesapeake Urology Research Assoc., Towson, Maryland
  - Five Valleys Urology, Missoula, Montana
  - Urological Institute of NE New York, Albany, New York
  - AMP of NY, Oneida, New York
  - AMP of NY, Syracuse, New York
  - Carolina Clinical Trials, Concord, North Carolina
  - The Urology Group, Cincinnati, Ohio
  - UCSEPA, Bala-Cynwyd, Pennsylvania
  - West Clinic, Memphis, Tennessee
  - Urology of Virginia, Virginia Beach, Virginia
  - Seattle Cancer Care Alliance, Univ. of Washington, Seattle, Washington

REFERENCES:
- [Derived] Yu EY, Getzenberg RH, Coss CC, Gittelman MM, Keane T, Tutrone R, Belkoff L, Given R, Bass J, Chu F, Gambla M, Gaylis F, Bailen J, Hancock ML, Smith J, Dalton JT, Steiner MS. Selective estrogen receptor alpha agonist GTx-758 decreases testosterone with reduced side effects of androgen deprivation therapy in men with advanced prostate cancer. Eur Urol. 2015 Feb;67(2):334-41. doi: 10.1016/j.eururo.2014.06.011. Epub 2014 Jun 24. PMID 24968970

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GTx-758 125mg | GTx-758 250 mg
Started | 38 | 39
Completed | 23 | 19
Not Completed | 15 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GTx-758 125mg | GTx-758 250 mg | Total
Number analyzed (Participants) | 38 | 39 | 77
Age, Continuous [Median (Full Range); unit: years] | 71 [51 to 88] | 69 [55 to 91] | 70 [51 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 38 | 39 | 77
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 33 | 34 | 67
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 33 | 21 | 54
  Hungary | 5 | 18 | 23

OUTCOME MEASURES:

1. Primary Outcome: Decline in Serum PSA
Description: The percentage of subjects with a 50% decline from baseline in serum PSA (confirmed by a second serum PSA assessment 30 days later) by Day 90 (with follow up confirmation by Day 120)
Time Frame: 120 days
Measure: Number; unit: participants
Arm/Group | GTx-758 125mg | GTx-758 250 mg
Number analyzed (Participants) | 38 | 39
participants | 4 | 10

ADVERSE EVENTS:
Time Frame: From time of screening to end of study, up to 4 years
Arm/Group | GTx-758 125mg | GTx-758 250 mg
All-Cause Mortality (participants affected / at risk) | 1/38 | 1/39
Serious Adverse Events (participants affected / at risk) | 1/38 | 10/39
Other Adverse Events (participants affected / at risk) | 31/38 | 33/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GTx-758 125mg (N=38) | GTx-758 250 mg (N=39)
Acute pyelonephritis (Renal and urinary disorders) | 1 | 0
Urinary Tract Infection (Renal and urinary disorders) | 1 | 0
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
acute renal failure (Renal and urinary disorders) | 1 | 5
pulmonary embolism (Cardiac disorders) | 0 | 3
acute myocardial infarction (Cardiac disorders) | 0 | 3
venous thrombosis (Cardiac disorders) | 0 | 3
pulmonary artery stenosis (Cardiac disorders) | 0 | 5
dehydration (Renal and urinary disorders) | 0 | 5
paraplegia (Musculoskeletal and connective tissue disorders) | 0 | 5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GTx-758 125mg (N=38) | GTx-758 250 mg (N=39)
anemia (Blood and lymphatic system disorders) | 3 | 3
bruising (Blood and lymphatic system disorders) | 1 | 0
leukocytosis (Blood and lymphatic system disorders) | 0 | 1
lymph node calcification (Blood and lymphatic system disorders) | 1 | 0
acute coronary syndrome (Cardiac disorders) | 0 | 1
angina (Cardiac disorders) | 2 | 1
AV block, first degree (Cardiac disorders) | 2 | 1
bradycardia (Cardiac disorders) | 1 | 0
bundle branch block, right (Cardiac disorders) | 0 | 1
cardiac aneurysm (Cardiac disorders) | 1 | 0
congestive heart failure (Cardiac disorders) | 1 | 0
cardiomegaly (Cardiac disorders) | 1 | 0
coronary artery disease (Cardiac disorders) | 3 | 2
left ventricular hypertrophy (Cardiac disorders) | 1 | 0
myocardial infarction (Cardiac disorders) | 1 | 0
ventricular extrasystoles (Cardiac disorders) | 1 | 0
adenomatous polyposis coli (Congenital, familial and genetic disorders) | 0 | 1
asplenia (Congenital, familial and genetic disorders) | 0 | 1
deafness, bilateral (Ear and labyrinth disorders) | 0 | 1
deafness, neurosensory (Ear and labyrinth disorders) | 0 | 1
tinnitus (Ear and labyrinth disorders) | 1 | 2
vertigo (Ear and labyrinth disorders) | 1 | 0
adrenal mass (Endocrine disorders) | 1 | 0
goiter (Endocrine disorders) | 0 | 1
hyperthyroidism (Endocrine disorders) | 0 | 2
hypogonadism (Endocrine disorders) | 0 | 1
hypothyroidism (Endocrine disorders) | 4 | 1
cataracts (Eye disorders) | 1 | 1
glaucoma (Eye disorders) | 2 | 3
lacrimation increased (Eye disorders) | 1 | 0
visual impairment (Eye disorders) | 1 | 0
strabismus (Eye disorders) | 0 | 1
abdominal discomfort (Gastrointestinal disorders) | 0 | 1
abdominal hernia (Gastrointestinal disorders) | 1 | 0
abdominal pain (Gastrointestinal disorders) | 2 | 0
anal fissure (Gastrointestinal disorders) | 1 | 0
barrett's oesophagus (Gastrointestinal disorders) | 1 | 0
constipation (Gastrointestinal disorders) | 6 | 0
diverticulum (Gastrointestinal disorders) | 2 | 1
dysphagia (Gastrointestinal disorders) | 1 | 0
gastric ulcer (Gastrointestinal disorders) | 1 | 0
gastroesophageal reflux (Gastrointestinal disorders) | 8 | 8
haematochezia (Gastrointestinal disorders) | 0 | 1
hemorrhoids (Gastrointestinal disorders) | 1 | 2
hiatus hernia (Gastrointestinal disorders) | 1 | 0
inguinal hernia (Gastrointestinal disorders) | 4 | 0
intestinal cyst (Gastrointestinal disorders) | 1 | 0
irritable bowl syndrome (Gastrointestinal disorders) | 0 | 29
large intestine polyp (Gastrointestinal disorders) | 0 | 1
nausea (Gastrointestinal disorders) | 2 | 0
peptic ulcer (Gastrointestinal disorders) | 0 | 1
rectal stenosis (Gastrointestinal disorders) | 1 | 0
poor dental condition (Gastrointestinal disorders) | 1 | 0
vomiting (Gastrointestinal disorders) | 1 | 1
asthenia (General disorders) | 0 | 1
chest pain (General disorders) | 0 | 1
chills (General disorders) | 0 | 1
fatigue (General disorders) | 7 | 4
foaming at mouth (General disorders) | 1 | 0
oedema peripheral (General disorders) | 1 | 2
pain (General disorders) | 1 | 1
polyp (General disorders) | 1 | 0
xerosis (General disorders) | 0 | 1
cholelelithiasis (Hepatobiliary disorders) | 1 | 0
hepatic cyst (Hepatobiliary disorders) | 1 | 0
hepatic steatosis (Hepatobiliary disorders) | 1 | 0
allergy to venom (Immune system disorders) | 0 | 1
drug hypersensitivity (Immune system disorders) | 1 | 0
seasonal allergy (Immune system disorders) | 3 | 1
acarodermatitis (Infections and infestations) | 1 | 0
acute sinusitis (Infections and infestations) | 0 | 1
cystitis (Infections and infestations) | 0 | 1
diverticulitis (Infections and infestations) | 2 | 0
echinococciasis (Infections and infestations) | 0 | 1
fungal skin infection (Infections and infestations) | 1 | 0
herpes virus infection (Infections and infestations) | 1 | 0
herpes zoster (Infections and infestations) | 0 | 1
labyrinthitis (Infections and infestations) | 0 | 1
nasopharyngitis (Infections and infestations) | 0 | 1
sinusitis (Infections and infestations) | 1 | 1
upper respiratory tract infection (Infections and infestations) | 1 | 1
urinary tract infection (Infections and infestations) | 2 | 2
ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
back injury (Injury, poisoning and procedural complications) | 1 | 0
clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0
forearm fracture (Injury, poisoning and procedural complications) | 0 | 1
hip fracture (Injury, poisoning and procedural complications) | 1 | 0
humerus fracture (Injury, poisoning and procedural complications) | 2 | 1
infection related reaction (Injury, poisoning and procedural complications) | 1 | 0
jaw fracture (Injury, poisoning and procedural complications) | 1 | 0
joint injury (Injury, poisoning and procedural complications) | 1 | 0
limb injury (Injury, poisoning and procedural complications) | 0 | 2
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
rib fracture (Injury, poisoning and procedural complications) | 1 | 1
road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
skeletal injury (Injury, poisoning and procedural complications) | 0 | 1
spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
tendon rupture (Injury, poisoning and procedural complications) | 2 | 0
wrist fracture (Injury, poisoning and procedural complications) | 1 | 1
ARTHROSCOPY (Investigations) | 1 | 0
BLOOD CREATININE INCREASED (Investigations) | 0 | 1
BLOOD GLUCOSE INCREASED (Investigations) | 1 | 0
cardiac murmur (Investigations) | 1 | 0
COMPUTERISED TOMOGRAM ABNORMAL (Investigations) | 1 | 0
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 1 | 0
GLUCOSE URINE PRESENT (Investigations) | 1 | 0
HEART RATE IRREGULAR (Investigations) | 1 | 0
PROSTATE EXAMINATION ABNORMAL (Investigations) | 1 | 0
URINE KETONE BODY PRESENT (Investigations) | 1 | 0
VISUAL TRACKING TEST ABNORMAL (Investigations) | 1 | 0
WEIGHT DECREASED (Investigations) | 1 | 0
WEIGHT INCREASED (Investigations) | 0 | 2
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 | 2
DIABETES MELLITUS (Metabolism and nutrition disorders) | 2 | 4
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 11 | 6
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPERLIPIDAEMIA (Metabolism and nutrition disorders) | 5 | 5
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 0
IMPAIRED FASTING GLUCOSE (Metabolism and nutrition disorders) | 0 | 1
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 5 | 4
VITAMIN B12 DEFICIENCY (Metabolism and nutrition disorders) | 1 | 0
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 1 | 3
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 | 4
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 7 | 4
BACK PAIN (Metabolism and nutrition disorders) | 6 | 5
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 | 1
BURSITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
EXOSTOSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
INTERVERTEBRAL DISC DEGENERATION (Musculoskeletal and connective tissue disorders) | 1 | 2
INTERVERTEBRAL DISC DISORDER (Musculoskeletal and connective tissue disorders) | 0 | 1
JOINT RANGE OF MOTION DECREASED (Musculoskeletal and connective tissue disorders) | 1 | 0
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 1 | 0
JUVENILE IDIOPATHIC ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
KYPHOSCOLIOSIS (Musculoskeletal and connective tissue disorders) | 1 | 0
MOBILITY DECREASED (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 2 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 2 | 0
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 1 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 3 | 0
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 1
OSTEITIS DEFORMANS (Musculoskeletal and connective tissue disorders) | 1 | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 7 | 2
OSTEOPENIA (Musculoskeletal and connective tissue disorders) | 1 | 2
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 4 | 0
OSTEOSCLEROSIS (Musculoskeletal and connective tissue disorders) | 1 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 | 1
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 1 | 0
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 0 | 1
SPINAL DISORDER (Musculoskeletal and connective tissue disorders) | 1 | 0
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 1
SPONDYLITIS (Musculoskeletal and connective tissue disorders) | 2 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
LIPOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
MALIGNANT MELANOMA IN SITU (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
MESOTHELIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
METASTASES TO BONE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
DEMENTIA (Nervous system disorders) | 1 | 0
DIABETIC NEUROPATHY (Nervous system disorders) | 1 | 0
DIZZINESS (Nervous system disorders) | 1 | 0
DYSGEUSIA (Nervous system disorders) | 1 | 0
EPILEPSY (Nervous system disorders) | 0 | 1
ESSENTIAL TREMOR (Nervous system disorders) | 1 | 0
GUILLAIN-BARRE SYNDROME (Nervous system disorders) | 0 | 1
HEADACHE (Nervous system disorders) | 3 | 2
LETHARGY (Nervous system disorders) | 0 | 1
MIGRAINE (Nervous system disorders) | 1 | 1
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 | 5
PARAESTHESIA (Nervous system disorders) | 1 | 0
PIRIFORMIS SYNDROME (Nervous system disorders) | 0 | 1
RADICULOPATHY (Nervous system disorders) | 0 | 1
RESTLESS LEGS SYNDROME (Nervous system disorders) | 1 | 0
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 | 1
VERTEBROBASILAR INSUFFICIENCY (Nervous system disorders) | 0 | 1
ALCOHOL ABUSE (Psychiatric disorders) | 0 | 1
ANXIETY (Psychiatric disorders) | 3 | 3
CLAUSTROPHOBIA (Psychiatric disorders) | 0 | 1
DEPRESSION (Psychiatric disorders) | 6 | 4
DRUG ABUSE (Psychiatric disorders) | 0 | 1
INSOMNIA (Psychiatric disorders) | 6 | 5
LIBIDO DECREASED (Psychiatric disorders) | 1 | 0
MENTAL STATUS CHANGES (Psychiatric disorders) | 1 | 0
MIDDLE INSOMNIA (Psychiatric disorders) | 0 | 1
PSYCHOTIC DISORDER DUE TO GENERA MEDICAL CONDITION (Psychiatric disorders) | 1 | 0
BLADDER DIVERTICULUM (Renal and urinary disorders) | 1 | 0
BLADDER NECK OBSTRUCTION (Renal and urinary disorders) | 0 | 1
CHROMATURIA (Renal and urinary disorders) | 1 | 0
DYSURIA (Renal and urinary disorders) | 2 | 0
HAEMATURIA (Renal and urinary disorders) | 4 | 2
HYPERTONIC BLADDER (Renal and urinary disorders) | 2 | 0
HYDRONEPHROSIS (Renal and urinary disorders) | 2 | 0
LOWER URINARY TRACT SYMPTOMS (Renal and urinary disorders) | 0 | 2
MICTURITION URGENCY (Renal and urinary disorders) | 3 | 2
NEPHROLITHIASIS (Renal and urinary disorders) | 1 | 2
NOCTURIA (Renal and urinary disorders) | 14 | 3
POLLAKIURIA (Renal and urinary disorders) | 8 | 4
STRESS URINARY INCONTINENCE (Renal and urinary disorders) | 1 | 1
TERMINAL DRIBBLING (Renal and urinary disorders) | 2 | 0
URINARY HESITATION (Renal and urinary disorders) | 1 | 1
URINARY INCONTINENCE (Renal and urinary disorders) | 4 | 1
URINARY RETENTION (Renal and urinary disorders) | 2 | 1
URINE FLOW DECREASED (Renal and urinary disorders) | 1 | 1
URINE ODOUR ABNORMAL (Renal and urinary disorders) | 1 | 0
URETHRAL STENOSIS (Renal and urinary disorders) | 2 | 0
BALANITIS (Reproductive system and breast disorders) | 1 | 0
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 5 | 5
BREAST PAIN (Reproductive system and breast disorders) | 1 | 1
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 17 | 5
GYNAECOMASTIA (Reproductive system and breast disorders) | 3 | 1
PELVIC PAIN (Reproductive system and breast disorders) | 2 | 0
PROSTATE INDURATION (Reproductive system and breast disorders) | 0 | 1
PROSTATOMEGALY (Reproductive system and breast disorders) | 0 | 1
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 | 1
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 | 2
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PHARYNGEAL CYST (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PULMONARY GRANULOMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 3 | 1
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 2 | 0
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 3 | 1
UPPER-AIRWAY COUGH SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 1
ACTINIC KERATOSIS (Skin and subcutaneous tissue disorders) | 1 | 0
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 1 | 2
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 1 | 0
SOLAR DERMATITIS (Skin and subcutaneous tissue disorders) | 1 | 0
ABDOMINAL HERNIA REPAIR (Surgical and medical procedures) | 0 | 2
APPENDICECTOMY (Surgical and medical procedures) | 3 | 0
ARTIFICIAL URINARY SPHINCTER IMPLANT (Surgical and medical procedures) | 1 | 0
BLADDER CALCULUS REMOVAL (Surgical and medical procedures) | 1 | 0
BLADDER NEOPLASM SURGERY (Surgical and medical procedures) | 1 | 0
CATARACT OPERATION (Surgical and medical procedures) | 2 | 1
CHOLECYSTECTOMY (Surgical and medical procedures) | 4 | 2
CIRCUMCISION (Surgical and medical procedures) | 1 | 0
COLECTOMY (Surgical and medical procedures) | 1 | 0
CYST REMOVAL (Surgical and medical procedures) | 1 | 0
DEBRIDEMENT (Surgical and medical procedures) | 1 | 0
DUODENAL ULCER REPAIR (Surgical and medical procedures) | 1 | 0
FRACTURE TREATMENT (Surgical and medical procedures) | 1 | 1
GASTRIC ULCER SURGERY (Surgical and medical procedures) | 1 | 0
HAEMORRHOID OPERATION (Surgical and medical procedures) | 2 | 1
HERNIA REPAIR (Surgical and medical procedures) | 1 | 1 (1)
HIP SURGERY (Surgical and medical procedures) | 1 | 0
INGUINAL HERNIA REPAIR (Surgical and medical procedures) | 1 | 0
JOINT DISLOCATION REDUCTION (Surgical and medical procedures) | 0 | 1
KNEE OPERATION (Surgical and medical procedures) | 1 | 0
OPEN REDUCTION OF FRACTURE (Surgical and medical procedures) | 1 | 0
RETINAL OPERATION (Surgical and medical procedures) | 0 | 2
CHONDROPLASTY (Surgical and medical procedures) | 1 | 0
SKIN NEOPLASM EXCISION (Surgical and medical procedures) | 2 | 0
SPINAL FUSION SURGERY (Surgical and medical procedures) | 0 | 1
SPINAL LAMINECTOMY (Surgical and medical procedures) | 1 | 0
STENT PLACEMENT (Surgical and medical procedures) | 1 | 0
TENDON OPERATION (Surgical and medical procedures) | 1 | 0
THYROIDECTOMY (Surgical and medical procedures) | 0 | 2
TONSILLECTOMY (Surgical and medical procedures) | 3 | 3
TYMPANOPLASTY (Surgical and medical procedures) | 0 | 1
URETHROTOMY (Surgical and medical procedures) | 1 | 0
VARICOSE VEIN OPERATION (Surgical and medical procedures) | 0 | 1
VASECTOMY (Surgical and medical procedures) | 2 | 2
WISDOM TEETH REMOVAL (Surgical and medical procedures) | 1 | 0
AORTIC ANEURYSM (Surgical and medical procedures) | 2 | 0
AORTIC DISSECTION (Surgical and medical procedures) | 1 | 0
ARTERIOSCLEROSIS (Vascular disorders) | 1 | 1
EMBOLISM (Vascular disorders) | 1 | 0
HOT FLUSH (Vascular disorders) | 10 | 11
HYPERTENSION (Vascular disorders) | 24 | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No